CLINICAL TRIAL: NCT01013181
Title: Safety and Efficacy of Romiplostim in Immune Thrombocytopenia (ITP) in the " Real-life " : Result of the French Experience in 72 Adults
Acronym: ATU-r
Status: Completed | Type: Observational
Sponsor: Henri Mondor University Hospital (Other)
Collaborators: Amgen (Industry); Paris 12 Val de Marne University (Other)
Responsible Party: Amgen Laboratory, Amgen Laboratory
Other Study IDs: ATU Romiplostim registry
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2009-11-17 (Estimated); Status verified 2009-11

CONDITIONS: Thrombopenia
Keywords: Immune Thrombopenia; Thrombocytopenia; romiplostim; compassionate program
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to review the charts of the first 100 patients included in the french compassionate program including patients with Immune Thrombopenia receiving romiplostim.

DETAILED DESCRIPTION:
Inclusion Criteria:

* Subject has a diagnosis of ITP according to the American Society of Hematology guidelines (George et al., 1996).
* Subject is equal to or greater than 18 years of age.
* Before any study-specific procedure, the appropriate written informed consent must be obtained.
* Subject receiving romiplostim in the compassionate program
* Available follow-up of one-year

Exclusion Criteria:

•Secondary ITP e.g: thrombopenia related to hepatitis C, HIV, Chronic Lymphocytic Leukemia...

The goal of this study is to review retrospectively the charts of the 100 first patients including in this program in France during the period of January 2008 and July 2008.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  * Subject has a diagnosis of ITP according to the American Society of Hematology guidelines (George et al., 1996).
  * Subject is equal to or greater than 18 years of age.
  * Before any study-specific procedure, the appropriate written informed consent must be obtained.

Exclusion Criteria:

* Exclusion Criteria:

  * Secondary ITP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary Immune Thrombopenia receiving romiplostim in a compasionnate program
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Safety and Efficacy of Romiplostim in Immune Thrombocytopenia (ITP)

REFERENCES:
- [Derived] Khellaf M, Michel M, Quittet P, Viallard JF, Alexis M, Roudot-Thoraval F, Cheze S, Durand JM, Lefrere F, Galicier L, Lambotte O, Panelatti G, Slama B, Damaj G, Sebahoun G, Gyan E, Delbrel X, Dhedin N, Royer B, Schleinitz N, Rossi JF, Mahevas M, Languille L, Bierling P, Godeau B. Romiplostim safety and efficacy for immune thrombocytopenia in clinical practice: 2-year results of 72 adults in a romiplostim compassionate-use program. Blood. 2011 Oct 20;118(16):4338-45. doi: 10.1182/blood-2011-03-340166. Epub 2011 Aug 10. PMID 21832276